CLINICAL TRIAL: NCT04665999
Title: Glycemic Profiles And Insulin Delivery Across The Menstrual Cycle In Women With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Chiara Fabris, PhD, Primary Investigator, University of Virginia
Other Study IDs: 190046
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Menstrual Cycle; Continuous Glucose Monitor (CGM); Oral contraceptives; Free cycling
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Free-cycling females: Continuous glucose monitor (CGM) data will be collected for three (3) full menstrual cycles. At the end of data collection, data will be analyzed to track insulin sensitivity and glycemic variability changes across the menstrual cycle. Participants will be asked to record meals consumed and free-cycling females will be asked to confirm ovulation by means of study-provided ovulation kits. Participants will be asked to record dates of beginning of menses and ovulation. Participants will also be provide an activity tracker to wear during the duration of the trial.
  Interventions: Device: Continuous Glucose Monitor
- Females taking Monophasic contraception: Continuous glucose monitor (CGM) data will be collected for three (3) full menstrual cycles. At the end of data collection, data will be analyzed to track insulin sensitivity and glycemic variability changes across the menstrual cycle. Participants will be asked to record meals consumed and free-cycling females will be asked to confirm ovulation by means of study-provided ovulation kits. Participants will be asked to record dates of beginning of menses and ovulation. Participants will also be provide an activity tracker to wear during the duration of the trial.
  Interventions: Device: Continuous Glucose Monitor

INTERVENTIONS:
Device: Continuous Glucose Monitor — Data collection only

SUMMARY:
This is an observational study. Forty females with type 1 diabetes (age 18-40) using a continuous glucose monitor and an insulin pump will be enrolled for a 3-month data collection. Study participants will include free-cycling females and females following oral contraceptive therapy. All study appointments may be completed virtually.

DETAILED DESCRIPTION:
Females, age 18-40 y.o., diagnosed with type 1 diabetes and currently using an insulin pump, will be provided a study continuous glucose monitor (CGM) in order to collect 3 full menstrual cycle data within 180 days. Enrollment may last from 3-5 months. Study participants will include free-cycling females and females following oral contraceptive therapy. Study CGMs and activity trackers will be provided for the entire data collection period. During data collection, all participants will be asked to record meals consumed and free-cycling females will be asked to confirm ovulation by means of study-provided ovulation kits. The Clue app will be recommended to study participants to record dates of beginning of menses and ovulation (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 12 months
* Use of glucose sensor in the last 6 months
* Use of insulin pump in the last 6 months
* Age ≥18 to ≤40 years
* HbA1c ≤8.5% if measured at screening or available from historical medical report performed within the last 6 months; in absence of a valid HbA1c measurement, average blood glucose estimated from CGM data to be approximately 200 mg/dL or less
* Absence of perimenopausal/menopausal symptoms
* Willingness to keep track of beginning of menstrual cycle
* Willingness to keep track of ingested carbohydrates
* Willingness to not become pregnant during study participation
* Regularly menstruating (at least every month with no missed cycles)
* Only free-cycling participants: willingness to use ovulation kits to confirm ovulation
* Only participants under oral contraceptive therapy: use of monophasic pill, with 3 weeks of active pill and 1 week of placebo
* Willingness to use the study Dexcom G6 during the study
* Participants must have Internet access and a computer system that meets the requirements for uploading the study equipment

Exclusion Criteria:

* Pregnancy
* Hormonal birth control therapy except monophasic pill contraceptive
* Polycystic ovary syndrome (PCOS) diagnosis
* Current use of steroids
* Concurrent use of any non-insulin glucose-lowering agent (including GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas, metformin)
* Uncontrolled thyroid disease
* Active fertility treatment
* Concomitant disease or condition that may compromise patient safety or ability to follow the protocol including: planned or current dialysis treatment; moderate to advanced nephropathy; known or suspected allergy to medical grade adhesives.
* Severe hypoglycemia or diabetes ketoacidosis (DKA) in the previous 6 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Regularly menstruating females (at least every month with no missed cycles)
Study Population: Females between the ages of 18 and 40 with no signs of menopause either free cycling or taking a monophasic contraception.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity computed using a Kalman filter-base algorithm embedding a model of glucose-insulin dynamics. | 3 months
  Primary Variable

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Fabris, PhD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT04665999/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT04665999/ICF_001.pdf